CLINICAL TRIAL: NCT05788484
Title: A Phase 1 Dose-escalation and Expansion Study of the PD-1 x ILT4 Bispecific Antibody CDX-585 in Patients With Advanced Malignancies
Brief Title: A Study of CDX-585 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX585-01
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer; Gastric Cancer; Head and Neck Cancer; Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Bladder Urothelial Carcinoma; Colorectal Cancer; Esophageal Cancer; Hepatic Cancer; Renal Cell Carcinoma; Cholangiocarcinoma; Pancreatic Cancer; Other Solid Tumors
Keywords: LILRB2; CD85d; ILT-4; PD1; Bi-Specific; Immunotherapy; Solid tumor Malignancies; Dose escalation; Immunological
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Head and Neck Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Carcinoma, Renal Cell; Cholangiocarcinoma; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDX-585 (Experimental): Dose-escalation phase: Eligible patients will receive treatment, based on cohort assigned, in 2-week cycles until progression or intolerance.
  Expansion phase: Patients enrolled in the expansion phase of the study will receive CDX-585 at the dose level chosen during the escalation phase.
  Interventions: Drug: CDX-585

INTERVENTIONS:
Drug: CDX-585 — CDX-585 is administered by infusion every 2 weeks

SUMMARY:
This is an open-label, non-randomized, multicenter, dose-escalation and expansion study in patients with selected solid tumors.

DETAILED DESCRIPTION:
This study will determine the maximum tolerated dose of CDX-585 while also evaluating the safety, tolerability, and efficacy of CDX-585 in patients with cancer.

Eligible patients that enroll to the dose-escalation portion of the study will be assigned to one of several dose levels of CDX-585. The dose-escalation part of the study will test the safety profile of CDX-585 and determine which dose of CDX-585 will be studied in the expansion portions of the study.

All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

The expansion portion of the study will further evaluate the safety of CDX-585 in selected tumor types at the dose level chosen during the escalation part of the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Recurrent, locally advanced, or metastatic solid tumor cancer excluding primary central nervous system tumors (e.g., glioblastoma).
2. Receipt of standard therapy for the tumor type in the recurrent, locally advanced, or metastatic setting.
3. Measurable (target) disease by iRECIST.
4. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 3 months following last treatment.
5. Willingness to undergo a pre-treatment and on-treatment biopsy, if required.

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other monoclonal antibodies.
2. Previous treatment with any anti-ILT4 antibody.
3. Patients who have received more than 1 anti-PD-1 or anti-PD-L1 targeted therapy, including in the adjuvant setting.
4. Prior anti-PD-L1 based therapy within 12 weeks and prior anti-PD-1 based therapy within four weeks to the planned start of study treatment.
5. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers. For all other cancers, the patient must be disease-free for at least one year to be allowed to enroll.
6. Thrombotic events within the last six months prior to study treatment
7. Active, untreated central nervous system metastases.
8. Active autoimmune disease or documented history of autoimmune disease.
9. History of (non-infectious) pneumonitis or has current pneumonitis.

There are additional criteria your study doctor will review with you to confirm eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Dose escalation: To determine the maximum tolerated dose of CDX-585 and to select the CDX-585 dose(s) for evaluation in tumor-specific expansion cohorts | Approximately 12 months
  The rates of drug-related adverse events will be summarized, and maximum tolerated dose will be determined.
Tumor-specific expansion cohorts: To further evaluate the safety of CDX-585 by tumor type. | Approximately 6 months
  The rates of drug-related adverse events will be summarized, and further evaluated in specific tumor types.

SECONDARY OUTCOMES:
Safety and Tolerability of CDX-585 as assessed by CTCAE v5.0 | From first dose through 90 days after last dose
  The rates of drug-related adverse events will be summarized and evaluated.
Objective Response Rate | Assessed up to approximately 1-3 years.
  The percentage of patients who achieve a confirmed immune complete response (iCR) or immune partial response (iPR)
Clinical Benefit Rate | Assessed up to approximately 1-3 years.
  The percentage of patients who achieve best response of confirmed iCR or iPR, or immune stable disease (iSD) for at least four months
Duration of Response | First occurrence of a documented objective response to disease progression or death (up to approximately 1-3 years)
  The interval from which measurement criteria are first met for iCR or iPR until the first date that progressive disease is objectively documented
Progression-free Survival | Cycle 1, day 1 to the first occurrence of disease progression or death due to any cause (up to approximately 1-3 years)
  The time from start of study drug to time of progression or death, whichever occurs first
Overall Survival | The time from start of study drug to death from any cause (up to approximately 1-3 years)
  The time from start of study drug to death
Pharmacokinetic Evaluation | Prior to, during, and at multiple time points after doses 1-4. Prior to every other dose from fifth dose, and at 30 and 90 days post last dose of study treatment
  CDX-585 serum concentrations will be measured at specified visits
Immunogenicity Evaluation | Prior to the first three doses and every other dose from the fifth dose of study treatment, then 30 and 90 days after the last dose
  Samples will be obtained for assessment of human anti-CDX-585

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - George Washington University Cancer Center, Washington D.C., District of Columbia
  - AdventHealth Celebration, Celebration, Florida
  - Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Providence Cancer Institute, Portland, Oregon